CLINICAL TRIAL: NCT01399749
Title: A Comparative Clinical Trial for the Repair of Chondral Knee Defects: Transplantation of Autologous Cultured Chondrocytes vs. Autologous Mesenchymal Stem Cells Derived From Adipose Tissue
Brief Title: Autologous Mesenchymal Stem Cells vs. Chondrocytes for the Repair of Chondral Knee Defects
Acronym: ASCROD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz (Other)
Responsible Party: Alonso C. Moreno Garcia, La Paz University Hospital. Orthopedic Surgery and Traumatology Department
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLPTRA-2009-01; 2009-016628-29 (EudraCT Number)
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Articular Cartilage Lesion of the Femoral Condyle
Keywords: Cartilage; Articular; Femoral; Knee; Chondrocytes; Adipose tissue-derived mesenchymal stem cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous ASC implantation (Experimental): Treatment with autologous ASC
  Interventions: Other: Implantation of autologous cells
- Autologous Chondrocytes implantation (Active Comparator): Treatment with autologous chondrocytes
  Interventions: Other: Implantation of autologous cells

INTERVENTIONS:
Other: Implantation of autologous cells — Implantation of autologous ASC or chondrocytes, 1 million per cm² lesion, covered by autologous periosteal membrane
  Other Names: ACI

SUMMARY:
The objective of our study is to compare the safety and effectiveness of the use of autologous cultured adipose tissue-derived stem cells versus cultured autologous chondrocytes for the treatment of chondral knee lesions.

DETAILED DESCRIPTION:
Chondral knee lesions are frequent and produce important functional limitations and arthrosis development. Arthrosis is one of the most important causes of disability and its treatment with prosthetic surgery is associated with a high cost, and is not free of other complications. Several studies of cell therapy with autologous chondrocytes have shown efficacy in the treatment of this type of lesions, and currently is a common technique for the treatment of focal lesions of articular cartilage. Autologous chondrocyte transplant is associated with morbidity of the cartilage sample removal, which needs intra-articular surgery, and the limited tissue sample for culture. Adipose tissue-derived mesenchymal stem cells (ASC) have demonstrated chondrocytic differentiation and have been used in animal models for articular cartilage repair. Adipose tissue yields more ASC than chondrocytes are obtained from cartilage, and liposuction is simple and with less adverse events than arthroscopy. It is worth mentioned that culture conditions are less stringent for ASC than for chondrocytes, in terms of number of passages to obtain the amount of cells needed for implantation.

We propose a randomized clinical trial, in which we compare the surgical implantation of either autologous chondrocytes or autologous ASC to treat chondral knee lesions.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic focal articular cartilage lesion on the medial femoral condyle
* Lesion on femoral condyle between 1 and 5 cm²
* ICRS Grade III/IV
* Stable knee
* Signed patient informed consent

Exclusion Criteria:

* Clinically relevant member malalignment (> 5 degrees)
* Non stable knee
* Inflammatory joint disease
* Knee surgery in the last year (transplant, suture or resection of the meniscus, mosaicplasty, microfracture)
* Participation in concurrent trials or in the previous 3 months
* Subjects with hepatitis, HIV or syphilis
* Malignancy in the previous 5 years
* Alcohol and/or drug abuse
* Poor general health as judged by Investigator
* Clinically relevant second cartilage lesion on the patella
* Patellofemoral cartilage lesion
* Known allergy to gentamicin or penicillins (or presence of multiple severe allergies)
* Having received hyaluronic acid intra-articular injections in the affected knee within the last 6 months of baseline
* Taking specific OA drugs such as chondroitin sulfate, diacerein, n-glucosamine, piascledine, capsaicin within 2 weeks of the baseline visit
* Corticosteroid treatment by systemic or intra-articular route within the last month of baseline or intramuscular or oral corticosteroids within the last 2 weeks of baseline
* Chronic use of anticoagulants
* Uncontrolled diabetes
* Any concomitant painful or disabling disease of the spine,hips or lower limbs that would interfere with evaluation of the afflicted knee
* Any clinically significant or symptomatic vascular or neurologic disorder of the lower extremities
* Liver enzymes (SGOT, SGPT, Alkaline Phosphatase) of more then two times the upper limit of normal or any other result that is clinically important according to the Investigator
* CRP > 10 mg/l

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Hyaline cartilage production for chondral knee lesions repair | 18 months

SECONDARY OUTCOMES:
Efficacy: Clinical evolution | 18 months
  Changes in Clinical tests and SF-12 Health Survey over 18 months
Efficacy: Functional evolution | 18 months
  Changes in Western Ontario-McMaster Osteoarthritis Score(WOMAC) over 18 months
Efficacy: Functional evolution | 18 months
  Changes in Knee Society Score(KSS) over 18 months
Efficacy: Histological evaluation | 18 months
  Hyaline cartilage production by histological methods at 18 months
Efficacy: Radiological evaluation | 18 months
  MRI at 18 months
Safety: Adverse events | 18 months
  Sistemic and local AEs especially attributable to implanted cells
Safety: Acute inflammatory events | 18 months
  Increase of pain of at least 30 mm on a 100 mm visual analog scale (VAS) along with self-reported swelling within 3 days post-cell application

CONTACTS AND LOCATIONS:
Overall Officials: Alonso C. Moreno Garcia, MD, Principal Investigator — Orthopedic Surgery and Traumatology Department. Knee Unit
Locations (1):
- La Paz University Hospital. Orthopedic Surgery and Traumatology Department, Knee Unit; Cell Therapy Laboratory., Madrid, Madrid, Spain

REFERENCES:
- [Background] Brittberg M, Lindahl A, Nilsson A, Ohlsson C, Isaksson O, Peterson L. Treatment of deep cartilage defects in the knee with autologous chondrocyte transplantation. N Engl J Med. 1994 Oct 6;331(14):889-95. doi: 10.1056/NEJM199410063311401. PMID 8078550
- [Background] Wakitani S, Imoto K, Yamamoto T, Saito M, Murata N, Yoneda M. Human autologous culture expanded bone marrow mesenchymal cell transplantation for repair of cartilage defects in osteoarthritic knees. Osteoarthritis Cartilage. 2002 Mar;10(3):199-206. doi: 10.1053/joca.2001.0504. PMID 11869080
- [Background] Garcia-Gomez I, Elvira G, Zapata AG, Lamana ML, Ramirez M, Castro JG, Arranz MG, Vicente A, Bueren J, Garcia-Olmo D. Mesenchymal stem cells: biological properties and clinical applications. Expert Opin Biol Ther. 2010 Oct;10(10):1453-68. doi: 10.1517/14712598.2010.519333. PMID 20831449